CLINICAL TRIAL: NCT05985187
Title: A Multicenter, Randomized, Double-blind, Parallel-controlled Clinical Study to Evaluate the Efficacy and Safety of TQB2440 Injection/Perjeta ® Combined With Trastuzumab and Docetaxel in Patients With Early or Locally Advanced ER/ PR-negative HER2-positive Breast Cancer.
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of TQB2440 Injection/Perjeta® Combined With Trastuzumab and Docetaxel in the Treatment of Patients With Early or Locally Advanced Breast Cancer.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB2440-III-01
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-04

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Trastuzumab; Docetaxel; pertuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2440 injection + Trastuzumab + docetaxel (Experimental): Neoadjuvant phase (cycle 1-4):
  TQB2440 injection + Trastuzumab + Docetaxel, intravenous infusion on the first day of each cycle, each cycle is 21 days.
  Adjuvant chemotherapy phase (cycle 5-7):
  Fluorouracil (600 mg/m2)+Epirubicin (90 mg/m2)+Cyclophosphamide (600mg/m2), intravenous injection once a day, on the first day of each cycle, each cycle is 21 days.
  Double targeted maintenance phase (cycle 8-20):
  TQB2440 injection+Trastuzumab, intravenous infusion on the first day of each cycle, each cycle is 21 days.
  Interventions: Drug: TQB2440 injection + Trastuzumab + Docetaxel
- Perjeta® + Trastuzumab + docetaxel (Active Comparator): Neoadjuvant phase (cycle 1-4):
  Perjeta® (Pertuzumab injection) + Trastuzumab + Docetaxel, intravenous infusion on the first day of each cycle, each cycle is 21 days.
  Adjuvant chemotherapy phase (cycle 5-7):
  Fluorouracil (600 mg/m2)+Epirubicin (90 mg/m2)+Cyclophosphamide (600mg/m2), intravenous injection once a day, on the first day of each cycle, each cycle is 21 days.
  Double targeted maintenance phase (cycle 8-20):
  TQB2440 injection+Trastuzumab, intravenous infusion on the first day of each cycle, each cycle is 21 days.
  Interventions: Drug: Perjeta + Trastuzumab + Docetaxel

INTERVENTIONS:
Drug: TQB2440 injection + Trastuzumab + Docetaxel — TQB2440 injection is a biosimilar of Perjeta® (Pertuzumab injection) developed by Chia Tai Tianqing Pharmaceutical Group. Trastuzumab is a recombinant DNA-derived human IgG monoclonal antibody against P185 glycoprotein regulated by HER2 gene in cell nucleus. Docetaxel is a selective L-type calcium channel blocker.
  Fluorouracil + epirubicin + cyclophosphamide for 3 cycles is a routine chemotherapy method after neoadjuvant surgery for breast cancer.
  The combination of Pertuzumab and Trastuzumab will enhance the antitumor activity and is used as the double targeted maintenance.
  Arms: TQB2440 injection + Trastuzumab + docetaxel
Drug: Perjeta + Trastuzumab + Docetaxel — Perjeta® with the general name Pertuzumab injection, is a recombinant humanized monoclonal antibody targeting the extracellular second domain of human epidermal growth factor receptor 2 (HER2). Trastuzumab is a recombinant DNA-derived human IgG monoclonal antibody against P185 glycoprotein regulated by HER2 gene in cell nucleus. Docetaxel is a selective L-type calcium channel blocker.
  Fluorouracil + epirubicin + cyclophosphamide for 3 cycles is a routine chemotherapy method after neoadjuvant surgery for breast cancer.
  The combination of Pertuzumab and Trastuzumab will enhance the antitumor activity and is used as the double targeted maintenance.
  Arms: Perjeta® + Trastuzumab + docetaxel

SUMMARY:
This is a multicenter, randomized, double-blind, parallel-controlled Phase III study to evaluate the efficacy and safety of TQB2440 injection/Perjeta® combined with trastuzumab and docetaxel in patients with early or locally advanced ER/ PR-negative HER2-positive breast cancer. The trial is scheduled to enroll 412 participants. The sample size was estimated based on 20 treatment cycles and 6 recurrence visits.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed the informed consent, and the compliance was good;
* Age: 18-75 years old (when signing the informed consent form); Eastern Cooperative Oncology Group Physical condition scoring criteria score: 0-1; Survival is expected to exceed 3 months;
* Patients with primary breast cancer confirmed by histopathology or cytology；
* Primary tumor diameter > 2 cm measured by local standard assessment method, or lymph node positive lesions confirmed by clinical or imaging examination;
* The investigators determined that this was consistent with the American Joint Committee on Cancer (AJCC) 8th Edition of breast cancer Tumor Node Metastasis stage II-III C (T2-T4 plus any N, or any T plus N1-3, M0) and histologically proven invasive breast cancer. A patient with invasive breast cancer must have a solid lesion capable of coarse needle biopsy;
* Laboratory tests confirmed HER2 positive, defined as a 3+ immunohistochemical result or a positive Fluorescence in situ hybridization double probe (2018 edition of American Society of Clinical Oncology/College of American Pathologists HER2 Testing Guidelines)
* The confirmed estrogen receptor (ER) and progesterone receptor (PgR) were negative;
* The patient agrees to undergo a mastectomy when surgical criteria are met after neoadjuvant therapy;
* Major organs function well, meeting the following criteria:

  1. Blood routine test criteria (no blood transfusion within 7 days prior to screening, no hematopoietic stimulant drug correction):

     1. Hemoglobin (HGB) ≥90g/L;
     2. Neutrophil absolute value (NEUT) ≥1.5×10^9/L;
     3. Platelet count (PLT) ≥ 100×10^9/L;
     4. Leukocyte ≥2.5×10^9/L;
  2. Biochemical tests must meet the following criteria:

     1. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN);
     2. Alanine transferase (ALT) and aspartate transferase (AST) ≤ 1.5×ULN.
     3. Serum creatinine (CR) ≤1.5×ULN or creatinine clearance (CCR) ≥50 ml/min (creatinine clearance calculated according to Cockcroft-Gault formula);
  3. The coagulation function test should meet the following criteria:

     1. Prothrombin time (PT), activated partial thromboplastin time (APTT), International Normalized ratio (INR) ≤ 1.5×ULN (no anticoagulant therapy), if the patient is receiving anticoagulant therapy, as long as the PT is within the intended range of anticoagulant drug use;
* For women who are not menopausal (menopause is defined as non-treaty-induced menopause for ≥12 months) or who are not surgically sterilized (removal of ovaries and/or uterus): Consent is required to remain abstinent during treatment and for at least 7 months after the last study treatment, or to take a single or combined annual failure rate of < 1% of non-hormonal contraception;
* For women of childbearing age, premenopausal or postmenopausal abstinence of less than 12 months, and who have not been surgically sterilized, serological pregnancy tests are negative.

Exclusion Criteria:

* Patients with stage IV metastatic breast cancer or other cancers that investigators determined could not be radically removed by neoadjuvant therapy;
* Bilateral invasive breast cancer;
* Patients with breast cancer who have previously received anti-tumor therapy, such as chemotherapy, endocrine therapy or anti-HER2 biotherapy, or who have undergone breast surgery (other than diagnostic biopsies for primary breast cancer);
* Occurred or present with other malignant tumors within 3 years. Patients with the following two conditions can be enrolled: other malignancies treated with a single operation, achieving continuous 5-year disease-free survival (DFS); Cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (cancer in situ) and T1 (tumor infiltrating basal membrane)];
* Major surgical treatment, open biopsy, or significant traumatic injury (except for diagnostic biopsies for primary breast cancer) received within 28 days before the start of study treatment;
* A wound or fracture that has not healed for a long time.
* Arteriovenous thrombosis occurred within 6 months, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
* Subject who have a history of psychotropic substance abuse and are unable to abstain or have mental disorders;
* Subjects with any severe and/or uncontrolled disease, including:

  1. Patients with a history of critical hypertension or hypertensive encephalopathy; Or uncontrolled high blood pressure (systolic blood pressure >150 mmHg after taking antihypertensive drugs, or diastolic blood pressure >100 mmHg);
  2. Heart failure or systolic dysfunction (LVEF < 55%) diagnosis history;
  3. Have grade 2 myocardial ischemia or myocardial infarction, arrhythmia (including QTc ≥450 ms in men, QTc ≥470 ms in women, and grade 2 congestive heart failure (NYHA rating);
  4. Angina pectoris requiring treatment with anti-angina medication;
  5. Valvular heart disease of clinical significance;
  6. Screening period confirmed hepatitis C virus (HCV) positive, human immunodeficiency virus (HIV) positive, syphilis treponema specific antibody positive, HBsAg positive and peripheral blood hepatitis B virus DNA (HBV DNA) titer beyond the normal range;
* Within 2 weeks before the start of the study treatment, the patients were treated with Chinese patent medicines (including compound Cantharides capsule, Kangai injection, Kanglaite capsule/injection, Aidi injection, Brucea javanica oil injection/capsule, Xiaoaiping tablet/injection, Cinobufacini capsule, etc.) which had clear anti-tumor indications in the China National Medicinal Products Administration (NMPA) approved drug label;
* Patients whose imaging (Computed Tomography or Magnetic Resonance Imaging) shows that the tumor has invaded an important blood vessel or who are judged by the investigator to be highly likely to invade an important blood vessel during subsequent studies and cause a fatal hemorrhage;
* Active autoimmune disease requiring systemic treatment (such as use of disease-modifying drugs, corticosteroids, or immunosuppressants) occurred within 2 years prior to study treatment initiation. Replacement therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic;
* Subjects diagnosed with immune deficiency or is receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy. (Dose >10mg/ day of prednisone or other therapeutic hormone) and continued use within 2 weeks of initial administration;
* Other comorbidities that interfere with planned treatment include severe lung dysfunction/disease, active or uncontrolled severe infection (≥ Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 grade 2 infection)
* Allergy to any investigational drug or any ingredient or excipient in the drug;
* Subjects had participated in clinical trials of other antineoplastic drugs within 4 weeks before the group;
* Participants who, in the investigator's judgment, have a concomitant medical condition that seriously endangers the safety of the subjects or interferes with the completion of the study, or who are deemed unsuitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-01-08 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Overall pathological complete response (tpCR) rate assessed by Independent review committee (IRC). | Baseline up to 4 months.
  Percentage of subjects with tumor shrinkage reached a complete response assessed by the IRC, defined as no invasive tumor cells in breast and axilla after primary tumor resection.

SECONDARY OUTCOMES:
tpCR rate evaluated by the investigators. | Baseline up to 4 months.
  Percentage of subjects with tumor shrinkage reached a complete response assessed by the investigators, defined as no invasive tumor cells in breast and axilla after primary tumor resection.
Breast pathological complete response (bpCR) rate evaluated by the investigators. | Baseline up to 4 months.
  It is defined as no invasive tumor cells in breast examined by microscopy after primary tumor resection, as assessed by the investigators.
bpCR assessed by IRC. | Baseline up to 4 months.
  It is defined as no invasive tumor cells in breast examined by microscopy after primary tumor resection, as assessed by the IRC.
Breast conservation rate | Baseline up to 5 months.
  Proportion of patients undergoing breast preservation surgery.
Objective remission rate (ORR) | Baseline up to 2 years.
  The optimal ORR evaluated by the investigator, including cases with complete response (CR) and partial response (PR).
Event-free survival (EFS) | Baseline up to two years.
  EFS refers to the time interval from randomization to the first recording of the following events: Preoperative disease progression as measured by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Disease free survival (DFS) | Baseline up to 2 years.
  DFS refers to the interval between the first day of absence of disease and the first recording of postoperative recurrence of disease or death from any cause, whichever comes first.
Overall Survival (OS) | Baseline up to 2 years.
  OS indicates the time interval from randomization to death from any cause.
Incidence of adverse events | Baseline up to 2 years.
  It refer to all adverse medical events that occur after patients or subjects receives an investigational drug, including adverse events (AE), serious adverse events (SAE), and treatment-related adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Sun Yat-sen University Cancer Prevention Center, Guangzhou, Guangdong
  - Affiliated cancer hospital of harbin medical university, Harbin, Heilongjiang
  - The First Affiliated Hospital of PLA Air Force Medical University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Xu D, Wu J, Yu J, Yang Y, Wen X, Yang J, Wei H, Xu X, Li Y, Yang L, Wang L, Wang Y, Ma W, Li N. A historical controlled study of domestic trastuzumab and pertuzumab in combination with docetaxel for the neoadjuvant treatment of early HER2-positive breast cancer. Front Oncol. 2024 Feb 9;14:1281643. doi: 10.3389/fonc.2024.1281643. eCollection 2024. PMID 38406813